CLINICAL TRIAL: NCT04765176
Title: A European Post-Market Clinical Follow-up Study (PMCF) in Patients With Infrarenal Aortic Aneurysm Undergoing Endovascular Stenting With the E-tegra Stent Graft System
Brief Title: A PMCF Study in Patients With Infrarenal Aortic Aneurysm Treated With the E-tegra Stent Graft System
Acronym: EASY
Status: Active, not recruiting | Type: Observational
Sponsor: JOTEC GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: EASY
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Vascular Aneurysm
Keywords: Abdominal; Aorta; Aneurysm; Endovascular; Repair
MeSH Terms: conditions — Aneurysm | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Endovascular Repair — Endovascular repair of the infrarenal aorta using a AAA stent graft.

SUMMARY:
The EASY post-market clinical follow-up study is undertaken to demonstrate safety and clinical performance of the E-tegra Stent Graft System used in endovascular treatment of infrarenal aortic aneurysm.

DETAILED DESCRIPTION:
In this study, patients will be observed who receive an E-tegra Stent Graft for the treatment of infrarenal aortic aneurysm. The E-tegra Stent Graft will be implanted at the discretion of the treating physician.

Participating physicians will provide their observations collected during routine care for patients they have decided to treat with the E-tegra stent graft. Informed consent of the patients to the use of their clinical records for study purposes will be obtained before their data will be collected in the post-market clinical follow-up study. All patients will be asked to complete questionaires focussing on the health status (HS) (SF-12) and Quality of Life (QoL) (WHOQOL-BREF).

The period of data collection will be approximately 60 months from the date of intervention for each patient. Source document verification will be performed on 100% of the patients; data from all visits will be reviewed and verified against existing source documents. Complete DICOM image files of the CT scans as well as other imaging files (e.g. CEUS, MRT) will be sent to a CoreLab for independent second evaluation. There is no CoreLab screening before inclusion. All adverse events defined prior to study start, will be adjudicated by the Clinical Evaluation Committee (CEC).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Patient must have an infrarenal aortic aneurysm with diameter ≥ 50 mm in females and ≥ 55 mm in males, or infrarenal aortic aneurysm with 40-50 mm that has increased in size by ≥ 1 cm per year
* Patient is elegible for treatment inside the instructions for use of the E-tegra Stent Graft System
* Patient is able and willing to undergo follow-up imaging and examinations prior to discharge from the hospital, at 30 days and 12 months, and annually thereafter until 5 years follow-up
* Patient understands and has signed the Informed Consent Form prior to intervention
* Patient has a life expectancy of at least 5 years

Exclusion Criteria:

* Patient with severe calcification or thrombi in the proximal sealing zone
* Patient with infectious aneurysm
* Patient with inflammatory aneurysm
* Patient with pseudoaneurysm
* Patient with symptomatic aneurysm
* Patient with ruptured or traumatic aneurysm
* Patient with suprarenal, juxtarenal, or pararenal aneurysm
* Patient with aortic dissection
* Patient with a reversed conical neck that is defined as a > 3 mm distal increase over a 15 mm length
* Patient in which the E-tegra Stent Graft System is used in combination with proximal or distal extenders of another company.
* Patient who is planned to be treated with an adjunctive aortic bare metal stent or a fenestrated stent graft
* Patient who is planned to be treated with a chimney / chimneys in the renal or visceral vessels
* Patient who is planned to be treated with an iliac branch device or parallel grafts in the iliac vessels
* Patient with genetic connective tissue disease (e.g. Marfan syndrome or Ehlers-Danlos syndrome)
* Patient with eGFR < 45 ml/min/1.73 m2 before the intervention
* Patient had or planned to have a major surgical or interventional procedure within 30 days before or 30 days after the planned implantation of the E-tegra Stent Graft System
* Patient with other medical condition that may cause the patient to be non-compliant with the protocol, confound the results, or is associated with a limited life expectancy of less than five years (i.e. heart failure, active malignancy (progressive, stable or partial remission))
* Patient who has been enrolled in another active clinical trial that does not allow inclusion in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients with asymptomatic infrarenal aortic aneurysm who are eligible for the endovascular treatment with the E-tegra Stent Graft System in accordance to the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30-day
  Rate of all-cause mortality

SECONDARY OUTCOMES:
Mortality | 24 hours, 12, 24, 36, 60 months
  Rate of all-cause mortality
Aneurysm-related mortality | 30-day, 12, 24, 36, 60 months
  Rate of aneurysm-related mortality
Aneurysm rupture-related mortality | 30-day, 12, 24, 36, 60 months
  Rate of aneurysm rupture-related mortality
Technical success | 24 hours
  Rate of patients with device technical success
Clinical success | 12 months
  Rate of patients with clinical success
Reintervention | 30-day, 12, 24, 36, 60 months
  Rate of patients with any reintervention
Reintervention-free survival | 12 months
  Rate of patients with reintervention-free survival
Primary limb patency | 30-day, 12, 24, 36, 60 months
  Rate of patients with primary E-tegra Stent Graft limb patency
Secondary limb patency | 30-day, 12, 24, 36, 60 months
  Rate of patients with secondary E-tegra Stent Graft limb patency
Stable aneurysm size | 12, 60 months
  Rate of patients with stable aneurysm size
Decreasing aneurysm size | 12, 60 months
  Rate of patients with decreasing aneurysm size on CTA scan (≤ 5 mm in maximum diameter)
Increasing aneurysm size | 12, 60 months
  Rate of patients with aneurysm growth on CTA scan (≥ 5 mm in maximum diameter)
Major adverse events | 30-day, 12, 24, 36, 60 months
  Rate of patients with major adverse events (aneurysm-related death, aneurysm rupture, new myocardial infarction requiring intervention (percutaneous transluminal coronary angioplasty, bypass), new disabling stroke (mRS ≥ 2), visceral ischemia (bowel ischemia with surgical/endovascular intervention or submission to ICU or bowel necrosis with surgical/endovascular intervention or submission to ICU), new hepatic infarction, new chronic (> 90 days) renal insufficiency/renal failure requiring dialysis, new permanent (> 30 days) paraplegia (modified Tarlov Scale ≤ 2), new permanent (> 30 days) paraparesis (modified Tarlov Scale 3 or 4), lower limb ischemia (increase in Rutherford classification)
Endoleak Type Ia | 12, 60 months
  Rate of patients with Type Ia endoleak
Endoleak Type Ib | 12, 60 months
  Rate of patients with Type Ib endoleak
Endoleak Type II | 12, 60 months
  Rate of patients with Type II endoleak
Endoleak Type III | 12, 60 months
  Rate of patients with Type III endoleak
Endoleak Type IV | 12, 60 months
  Rate of patients with Type IV endoleak
Endoleak of unknown origin | 12, 60 months
  Rate of patients with endoleak of unknown origin
Stent graft migration | 12, 60 months
  Rate of patients with stent graft migration > 10 mm
Dislodgement | 30-day, 12, 24, 36, 60 months
  Rate of patients with stent graft dislodgement (full component separation)
Stent fracture | 12, 60 months
  Rate of patients with stent fracture
Stent graft infection | 30-day, 12, 24, 36, 60 months
  Rate of patients with stent graft infection
Health status | 6, 12, 48 to 60 months
  Rate of patients with the same level of health status as prior to surgery
QoL | 6, 12, 48 to 60 months
  Rate of patients with the same level of QoL as prior to surgery

CONTACTS AND LOCATIONS:
Overall Officials: Michel MP Reijnen, Prof., Principal Investigator — Rijnstate
Locations (1):
- Rijnstate Hospital, Arnhem, Netherlands